CLINICAL TRIAL: NCT03599765
Title: External Beam Radiation to Eliminate Nominal Metastatic Disease (EXTEND): A Randomized Phase II Basket Trial Assessing the Efficacy of Upfront Local Consolidative Therapy (LCT) for Oligometastatic Disease
Brief Title: Systemic Therapy With or Without Local Consolidative Therapy in Treating Patients With Oligometastatic Solid Tumor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0349; NCI-2018-01469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0349 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Oligometastatic Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (LCT, routine therapy) (Experimental): Patients receive up-front standard of care LCT including but not limited to surgical resection, cryotherapy, and radiofrequency ablation. Patients then receive routine drug therapy.
  Interventions: Other: Best Practice; Procedure: Local Consolidation Therapy
- Arm II (routine therapy) (Experimental): Patients receive routine drug therapy. Patients may later receive LCT at the discretion of doctor.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive routine therapy
  Other Names: standard of care; standard therapy
Procedure: Local Consolidation Therapy — Receive LCT
  Other Names: LCT; Local Consolidative Therapy
  Arms: Arm I (LCT, routine therapy)

SUMMARY:
This phase II trial studies how well systemic therapy with or without local consolidative therapy work in treating patients with solid tumor that has spread to 1 site of other places in the body. Treatment with up-front local consolidative therapy may be better in helping to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In patients with oligometastatic malignancies, to assess PFS with upfront LCT vs. no LCT among randomized patients. In this analysis each disease site will be analyzed separately.

SECONDARY OBJECTIVES:

I. In patients with oligometastatic malignancies, to assess OS with upfront LCT vs. no LCT among randomized patients. In this analysis disease sites will be amalgamated and analysis will compare randomized arms.

II. In patients with oligometastatic malignancies, to assess time to next line systemic therapy with upfront LCT vs. no LCT. The subsequent line of systemic therapy will be defined as the subsequent line after protocol specified systemic therapy.

III. In patients with oligometastatic malignancies, to assess time to new lesion failure with upfront LCT vs. no LCT.

IV. To assess safety/tolerability of upfront LCT in patients with oligometastatic malignancies.

V. In patients with oligometastatic malignancies, to assess quality of life with upfront LCT vs. no LCT. Separate analyses will assess 1) all disease sites amalgamated and 2) all disease sites analyzed separately.

VI. In patients with oligometastatic malignancies, assess time to local failure with upfront LCT vs no LCT.

VII. In patients with oligometastatic prostate cancer, assess radiographic progression-free survival with upfront LCT vs no LCT. VIII. In patients with oligometastatic castrate-sensitive prostate cancer, assess castrateresistance free survival with upfront LCT vs no LCT.

EXPLORATORY OBJECTIVES:

I. To identify predictive/prognostic biomarkers that are associated with a benefit to LCT across disease sites.

II. To investigate alterations in biomarker profile over time and in response to radiation delivery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive up-front standard of care LCT including but not limited to surgical resection, cryotherapy, and radiofrequency ablation. Patients then receive routine drug therapy.

ARM II: Patients receive routine drug therapy. Patients may later receive LCT at the discretion of doctor.

After completion of study, patients are followed up every 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic solid tumors (see protocol for relevant disease sites) patients (=< 5 metastatic lesions at the time of study entry)
* Candidate for definitive local therapy to all sites of active disease per the discretion of the treating physicians
* No more than 4 prior lines of systemic therapy administered to treat metastatic disease
* Pathologically confirmed diagnosis of cancer as specified in protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 500/mcL (performed within 6 weeks prior to study enrollment)
* Platelets >= 25,000/mcL (performed within 6 weeks prior to study enrollment)
* Hemoglobin >=7 g/dL (performed within 6 weeks prior to study enrollment)
* Serum total bilirubin =< 1.5 mg/dl (except for subjects with Gilbert syndrome, who may have total bilirubin < 3.0 mg/dl) OR direct bilirubin =< upper limit normal (ULN) for subjects with total bilirubin levels > 1.5 mg/dl (performed within 6 weeks prior to study enrollment)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 3 X ULN OR =< 5 X ULN for subjects with liver metastases (performed within 6 weeks prior to study enrollment)

Exclusion Criteria:

* Has a diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy
* Metastatic effusion (e.g. pleural effusion or ascites). Note that patients with an effusion that is too small to sample will be eligible for the trial
* Diffuse metastatic processes including leptomeningeal disease, diffuse bone marrow involvement, and peritoneal carcinomatous, which by the discretion of the treating physician cannot be treated definitively
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* In the event that a curative systemic option exists for metastatic disease from a given disease site. First-line metastatic patients (those patients who have had no prior lines of systemic therapy targeting their metastatic disease) are only eligible for enrollment if they have completed their curative systemic therapy per the judgment of the treating oncologist and have persistent disease
* Is pregnant or expecting to conceive within the projected duration of the trial at the screening visit

  * Female subject of childbearing potential should have a negative urine or serum pregnancy within 6 weeks prior to study registration up to the first fraction of radiation
  * Note: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Additional diagnosis of another primary malignancy outside of the malignancy being treated on trial that per the discretion of the treating physicians and investigational team offers a substantial risk to the patient's life (e.g. primary lung cancer definitively treated in the past 6 months would offer a significant risk to the patient's life, while a basal cell carcinoma treated with local excision would not)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year
  General descriptive statistics will be computed.
Progression free survival | Up to 1 year
Time to development of new distant metastases | Up to 1 year
Overall survival | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, Principal Investigator — M.D. Anderson Cancer Center
Locations (12):
- United States (12):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Queen's Medical Center, Honolulu, Hawaii
  - Community Health Center, Coldwater, Michigan
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Ludmir EB, Sherry AD, Fellman BM, Liu S, Bathala T, Haymaker C, Medina-Rosales MN, Reuben A, Holliday EB, Smith GL, Noticewala SS, Nicholas S, Price TR, Martin-Paulpeter RM, Perles LA, Lee SS, Lee MS, Smaglo BG, Huey RW, Willis J, Zhao D, Cohen L, Taniguchi CM, Koay EJ, Katz MHG, Wolff RA, Das P, Pant S, Koong AC, Tang C. Addition of Metastasis-Directed Therapy to Systemic Therapy for Oligometastatic Pancreatic Ductal Adenocarcinoma (EXTEND): A Multicenter, Randomized Phase II Trial. J Clin Oncol. 2024 Nov 10;42(32):3795-3805. doi: 10.1200/JCO.24.00081. Epub 2024 Aug 5. PMID 39102622
- [Derived] Tang C, Sherry AD, Haymaker C, Bathala T, Liu S, Fellman B, Cohen L, Aparicio A, Zurita AJ, Reuben A, Marmonti E, Chun SG, Reddy JP, Ghia A, McGuire S, Efstathiou E, Wang J, Wang J, Pilie P, Kovitz C, Du W, Simiele SJ, Kumar R, Borghero Y, Shi Z, Chapin B, Gomez D, Wistuba I, Corn PG. Addition of Metastasis-Directed Therapy to Intermittent Hormone Therapy for Oligometastatic Prostate Cancer: The EXTEND Phase 2 Randomized Clinical Trial. JAMA Oncol. 2023 Jun 1;9(6):825-834. doi: 10.1001/jamaoncol.2023.0161. PMID 37022702
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org